CLINICAL TRIAL: NCT04607473
Title: Comparison of ABUS and HHUS in Preoperative Evaluation of Patients With Early-stage Breast Cancers
Brief Title: ABUS for Early-stage Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ji Soo Choi, Assistant Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GRO-06-001
Record Dates: First submitted 2020-10-18; First posted 2020-10-29 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Early Stage Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABUS (Experimental): ABUS is performed by experienced technicians using a GE inveniaTM. Each breast is imaged in three views with an automated 15.4-cm 14-6-MHz linear- array transducer, which acquires up to 1000 two-dimensional images in the transverse plane, imaging the breast in three parts: the central (anteroposterior), lateral, and medial portions of the breast. To ensure inclusion of all breast tissue, particularly in participants with very large breasts, additional views are obtained as deemed necessary by the technician to cover the entirety of the breast.
  Interventions: Device: automated breast ultrasound (ABUS)

INTERVENTIONS:
Device: automated breast ultrasound (ABUS) — Both HHUS and ABUS will be performed on each patient for preoperative staging. Breast radiologists each independently will read HHUS and ABUS images obtained from one patient. The radiologists will be blinded to the findings of the other US mode.
  Other Names: hand-held ultrasound (HHUS)

SUMMARY:
While the role of automated breast ultrasound (ABUS) as an alternative to hand-held ultrasound (HHUS) in breast cancer screening has been established, the use of ABUS in preoperative evaluation of newly diagnosed breast cancer patients is still limited. This may be because axillary areas are not included in the scanning area of ABUS. Newly diagnosed breast cancer patients have undergone axillary US to predict axillary lymph node metastasis before surgery, in combination with preoperative breast US, in many institutions. However, recent studies have reported that sentinel lymph node biopsy alone is sufficient for diagnosis and treatment of axillae of patients with early-stage breast cancer, because the incidence of axillary lymph node metastasis is very low. Therefore, the clinical significance of preoperative axillary US is being lowered in patients with early-stage breast cancers. Thus, considering that coronal images provided by ABUS may be more advantageous for detection of multifocal or multicentric cancer, we hypothesized that ABUS could replace HHUS in preoperative staging of patients with early-stage breast cancers (clinical Tis, T1-2/N0 cancers) for whom preoperative axillary US is not necessary. The purpose of this study was to prospectively compare the diagnostic performances of ABUS and HHUS in preoperative evaluation of patients with early-stage breast cancers. This study will be conducted with institutional review board approval, and written informed consent will be obtained. From the Jan 2019 to Dec 2021, 675 patients diagnosed with early-stage breast cancer will be enrolled from the three institutions. Both ABUS and HHUS will be performed on each patient before surgery. Breast radiologists independently review ABUS and HHUS images. They detect all visible lesions and record the location and size of them. They characterize all detected lesions by using BI-RADS category. The primary object is to compare the diagnostic performance of ABUS and HHUS as preoperative staging tool in women with known breast cancers. The sensitivities and specificity of each US mode for the detection of breast cancers are calculated on a per-lesion basis. McNemar's test and Fisher's exact test are used to compare the sensitivities and PPVs for ABUS and HHUS. Significance testing on the lesion level and patient level is conducted using generalized estimating equations (GEEs) with a logit link and an independent working correlation structure to adjust the effect of clustering on radiologists and patients. GEEs are utilized to compare the sensitivities and PPVs for ABUS and HHUS. Diagnostic performance are assessed with receiver operating characteristics curve analysis. Area under the curves are calculated from both parametric and trapezoidal curve fitting. Agreements between tumor size measured by each US mode and pathologic the tumor size are analyzed with the intraclass correlation coefficient (ICC) and 95% Bland-Altman limits of agreement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early-stage breast cancer (clinical Tis, T1- T2 cancers are suspected on mammography at the time of diagnosis), without palpable nodes at physical examination (N0)
* Patients who schedule to undergo surgery and sentinel lymph node biopsy
* Patient's age between 25-69 years
* Patients who voluntarily agree to participate in this study

Exclusion Criteria:

* A history of previously treated breast cancers
* Patients who undergo excision biopsy for diagnosed breast cancer
* Pregnant or lactating women
* Patients who have breast implants

Ages: 25 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performances of ABUS and HHUS | 3 year
  The sensitivities and specificity of each US mode for the detection of breast cancers are calculated on a per-lesion basis

SECONDARY OUTCOMES:
Agreement between tumor size measurements | 3 year
  Agreement between tumor size measurements by ABUS and HHUS and pathologic tumor size

CONTACTS AND LOCATIONS:
Overall Officials: Ji Soo Choi, MD,PhD, Principal Investigator — Samsung Medical Center, Department of Radiology
Locations (3):
- South Korea (3):
  - Department of Radiology, Konkuk University Medical Center, Konkuk University School of Medicine, Seoul
  - Samsung Medical Center, Seoul
  - Department of Radiology Ewha womans university medical center, Seoul

IPD SHARING:
Plan to Share IPD: No